CLINICAL TRIAL: NCT06569251
Title: Adverse Neonatal Outcomes with a Shortened Clinical Regimen of Dexamethasone: Single-blind Randomized Clinical Trial: UNODEXA Trial
Brief Title: Adverse Neonatal Outcomes with a Shortened Clinical Regimen of Dexamethasone.
Acronym: UNODEXA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ricardo A Gutierrez Ramirez, MD, MSc, FACOG (Other)
Responsible Party: Sponsor-Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Research Coordinator for the Postgraduate Program in Gynecology and Obstetrics, Universidad Nacional Autonoma de Honduras
Organization: Universidad Nacional Autonoma de Honduras (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGO-UNAH-47-1-2024
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-08

CONDITIONS: Preterm Birth; Distress Respiratory Syndrome
Keywords: preterm birth; Dexamethasone
MeSH Terms: conditions — Premature Birth; Pulmonary Atelectasis | interventions — Dexamethasone; BID protein, human

STUDY DESIGN:
Intervention Model Description: Experimental. Single-blind, parallel-group, non-inferiority randomized clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Both the patient and the principal investigator will know the intervention, the data analyst researcher does not know the group to which the patients have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group intervention (shortened dexamethasone regimen) (Experimental): Dexamethasone 12 mg IM every day for 2 days. Total dose: 24 mg
  Interventions: Drug: Dexamethasone 12 mg QD
- Group control (conventional dexamethasone regimen) (Active Comparator): Dexamethasone 6 mg IM every 12 hours for 2 days. Total dose: 24 mg.
  Interventions: Drug: Dexamethasone 6 mg BID

INTERVENTIONS:
Drug: Dexamethasone 12 mg QD — Administration of dexamethasone to the mother as an inducer of fetal lung maturity. shortened scheme
  Arms: Group intervention (shortened dexamethasone regimen)
Drug: Dexamethasone 6 mg BID — Administration of dexamethasone to the mother as an inducer of fetal lung maturity. standard Scheme
  Arms: Group control (conventional dexamethasone regimen)

SUMMARY:
Respiratory morbidity, including respiratory distress syndrome (RDS), is a serious complication of preterm birth and the leading cause of early neonatal mortality and disability. The effects of antenatal corticosteroid administration on fetal lung maturation have been widely studied in order to counteract such adverse perinatal outcomes of preterm birth. The dexamethasone regimen will be evaluated at different administration frequencies, but at the same total dose. The hypothesis is: The type of dexamethasone regimen administered for fetal lung maturation influences the incidence of perinatal complications.

DETAILED DESCRIPTION:
Prematurity is a major obstacle to achieving goal 4 of the Millennium Development Goals, given its high contribution to neonatal mortality. The survival chances of premature babies vary significantly depending on where they are born. Preterm birth has remained the major contributor to neonatal morbidity and mortality worldwide, accounting for 70% of neonatal deaths.

As a management to reduce neonatal morbidity and mortality secondary to preterm birth, corticosteroid regimens have been established to accelerate fetal lung maturation. The reduction in perinatal complication rates has been widely observed, however, no differentiation has been observed between the incidence of complications according to the scheme applied.

Neonatal complications of preterm birth include respiratory distress syndrome, bronchopulmonary dysplasia, cystic periventricular leukomalacia, patent ductus arteriosus, sepsis, intraventricular hemorrhage, necrotizing enterocolitis, hypothermia, hypoglycemia, hyperbilirubinemia, and feeding difficulties. Long-term morbidity includes retinopathy of prematurity, neurodevelopmental impairment, and cerebral palsy. Of these, respiratory morbidity, including respiratory distress syndrome (RDS), is a serious complication of preterm birth and the leading cause of early neonatal mortality and disability.

Preterm birth rates are highest in low- and lower-middle-income countries (11.8% and 11.3% on average, respectively), while rates are lowest in upper-middle- and high-income countries ( 9.4% and 9.3%, respectively). More than 60% of all premature births worldwide occur in low-resource, high-fertility countries. In Honduras, a study carried out from 1998-2000 at the Maternal and Child Hospital by Portillo M. et al, reported a prevalence of preterm birth of 4.7% (1929 premature births out of 40,786 births).

Experimental. Single-blind, parallel-group, non-inferiority randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Delivery of a signed and dated informed consent form.
2. Declared willingness to comply with all study procedures and availability during the duration of the study.
3. Pregnant patient with 20 or more weeks of gestation determined by USG with clinically diagnosed threat of preterm labor (defined as uterine contractions with sufficient progressive frequency and intensity that allow dilation of the cervix before the 37th week of gestation).
4. Pregnant patient admitted and birth in the Maternal and Child Hospital, Labor and Delivery room. Part.
5. Delivery carried out at the Teaching Hospital.
6. Patient with a diagnosis of premature rupture of membranes under conservative management.
7. patient must know how to read and write
8. Possess a cell phone or some other means of communication.
9. Residing in the city of Tegucigalpa, Honduras.

Exclusion Criteria:

1. Patients under 18 years of age.
2. Patient with diagnosed psychiatric illnesses.
3. Pregnant patient with threat of preterm birth who is also diagnosed with preeclampsia with data of severity and intrauterine growth restriction.
4. Pregnant patient with threat of preterm birth who is also diagnosed with premature rupture of membranes.
5. Pregnant patient with threat of preterm birth who is also diagnosed con corioamnionitis.
6. Pregnant patient with threat of preterm birth who is also diagnosed with acute abdomen.
7. Major fetal malformations
8. Fetal death

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 68 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
neonatal complications | from the first intervention to Newborn discharge. on average less than 28 days
  Presence or absence of respiratory distress syndrome, necrotizing enterocolitis, intraventricular hemorrhage, cystic ventricular leukomalacia, or death after receiving any of the different antenatal corticosteroid regimens

SECONDARY OUTCOMES:
Maternal complications | rom the first intervention to birth. on average less than 28 days
  Signs of maternal or neonatal infection determined clinically and laboratory after administration of corticosteroids. Maternal hyperglycemia or arterial hypertension. Fetal hypoglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Gutierrez Ramirez, MD, MSc, Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogel JP, Chawanpaiboon S, Moller AB, Watananirun K, Bonet M, Lumbiganon P. The global epidemiology of preterm birth. Best Pract Res Clin Obstet Gynaecol. 2018 Oct;52:3-12. doi: 10.1016/j.bpobgyn.2018.04.003. Epub 2018 Apr 26. PMID 29779863
- [Background] Brownfoot FC, Gagliardi DI, Bain E, Middleton P, Crowther CA. Different corticosteroids and regimens for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2013 Aug 29;(8):CD006764. doi: 10.1002/14651858.CD006764.pub3. PMID 23990333
- [Background] Kastanek M, Frommlet F, Linsenmeier L, Helmer H. Influence of antenatal corticosteroid lung maturation on maternal inflammatory parameters. J Matern Fetal Neonatal Med. 2022 Mar;35(6):1210-1212. doi: 10.1080/14767058.2020.1743653. Epub 2020 Mar 31. PMID 32233700